CLINICAL TRIAL: NCT05235035
Title: The Effect of Sleep Misalignment on the Cognitive Empathetic Ability to Recognize Pain and to Evaluate the Pain Intensity in Others as Competence for Qualitative Care
Brief Title: PAIN Empathy Assessment in Sleep Deprived Emergency & Acute Care Clinicians
Acronym: PAIN-EASE
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, Principal Investigator, Claude Bernard University
Other Study IDs: PAIN-EASE
Record Dates: First submitted 2022-01-07; First posted 2022-02-10 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Empathy; Sleep; Pain
Keywords: cognitive empathy; health care professionals; pain recognition; pain assessment; sleep misalignment; quality of care
MeSH Terms: conditions — Pain | interventions — Shift Work Schedule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- health care professionals: Staff from the department of anesthesia and general resuscitation and thoracic cardiac pediatric with patient contact that regularly works in shifts including night shifts
  Interventions: Behavioral: Night shift work

INTERVENTIONS:
Behavioral: Night shift work — Subjects are exposed to irregular sleep and sleep misalignment due to hospital night shifts.

SUMMARY:
Cognitive Empathy is relevant in clinical practice and will be assessed based on the accuracy of pain recognition and the pain intensity evaluation in a computerised task using facial expressions. Repeated measures across day and night shifts will provide the basis to understand the impact of shift work on those abilities in health care professionals.

DETAILED DESCRIPTION:
Assessment and management of the pain patients experience is one of the key skills needed in the field of anesthesiology. The consideration of non-verbal cues is essential, especially the recognition of facial expressions. The human ability to recognize emotions in others depends on the capacity for empathy of an individual, specifically cognitive empathy. In the clinical context empathy is understood as a set of skills and competences rather than a character trait. It may therefore vary due to various parameters. Currently there is no research available on the influence of shift work on the human ability to recognize pain in facial expressions. However, work schedules that do not fit the natural circadian rhythm are known to alter the processing of emotions. In particular the ability to judge the intensity of an emotion is influenced. Therefore, the hypothesis of the present study will be, that shift work impairs the pain assessment performance of an individual. To test this hypothesis, the effect of shift work on the performance in recognizing and assessing pain intensity of faces by health care professionals in the anesthesia department will be assessed. A repeated measures assessment will be used.

ELIGIBILITY:
Exclusion criteria:

* refuse to participate
* not working night shifts
* no patient contact

Inclusion criteria:

* working day and night shifts
* health care professional with patient contact

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Care Professionals:
  Nurses, nursing assistants, child care nurses and volunteer doctors from the department of anesthesia and general resuscitation and thoracic cardiac pediatric
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Comparison of pain recognition accuracy during day or night | 1 day, 1 night
  Pain recognition ability measured as accuracy (percentage correct responses / total responses) when subliminally presented with faces of different emotions in a computerised task : 48 trials including 1/3 of painful stimuli and 2/3 of non-pain stimuli (other distractor emotions are happy, disgusted, sad, angry, surprised). Stimuli from Delaware Pain Database.
  The change of accuracy during a shift (baseline measure at beginning of shift, post measure after shift) is compared between a day shift and a night shift
Comparison in pain intensity on NPRS - numerical pain rating scale | 1 day, 1 night
  Pain assessment ability is measured as intensity rating on the common NPRS 11-point Likert scale of 0 - 10 (0 representing no pain and 10 indicating maximum pain) when consciously presented with faces (48 trials) showing pain in different intensity levels in a computerized task including neutral distractors.
  Stimuli from Delaware Pain Database. The change of intensity evaluation during a shift (baseline measure at beginning of shift, post measure after shift) is compared between a day shift and a night shift

SECONDARY OUTCOMES:
Prior Shift - Total Sleep Time in h compared between shift types | 1 day, 1 night
  Before any shift participants are asked to give information on their sleeping behavior within the last 72 hours. The Total Sleep Time (TST = time asleep in bed excluding sleep latency and nocturnal awakenings) will be accumulated.
Nap Time during Shift in h compared between shift types | 1 day, 1 night
  After any shift participants are asked to give information on their sleeping behavior during the course of the shift. The Total Sleep Time (time asleep in bed excluding sleep latency and nocturnal awakenings) will be accumulated.
Empathy - Jefferson Scale of Physician Empathy | 1 day
  Empathy assessment by Jefferson Scale of Physician Empathy (JSPE; Zenasni et al., 2012). It is a brief self-report scale of 20 items with a 7-point Likert scale, ranging from 1= strongly disagree to 7=strongly agree (average Score between 1 and 7). Higher scores are indicating a higher level of empathy.
Prior Shift Recovery Quality on 5 point Likert Scale compared between shift types | 1 day, 1 night
  Before any shift participants are asked to give information on their sleeping behavior within the last 72 hours which also includes the subjective evaluation of sleep quality, waking quality and form of the day on a five point likert scale (1 = very bad to 5 = very good). A composed score of these three evaluations will be created and compared according to shift type.
  ((average Sleep + average Wakening + average Form)/3)
Comparison of speed in pain recognition task as cognitive performance during day or night shift | 1 day, 1 night
  Reaction time during the subliminal pain recognition task as additional marker of cognitive performance. The change of reaction time during a shift (baseline measure at beginning of shift, post measure after shift) is compared between a day shift and a night shift
Health Care Professional Work Expertise in years | 1 day
  Self-reported years of work experience as a health care professional
Shift Work Expertise in years | 1 day
  Self-reported years of work experience in a shift work system

CONTACTS AND LOCATIONS:
Locations (1):
- Claude Bernard University, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czeisler CA, Pellegrini CA, Sade RM. Should sleep-deprived surgeons be prohibited from operating without patients' consent? Ann Thorac Surg. 2013 Feb;95(2):757-66. doi: 10.1016/j.athoracsur.2012.11.052. No abstract available. PMID 23336899
- [Background] Gelinas C, Fillion L, Puntillo KA, Viens C, Fortier M. Validation of the critical-care pain observation tool in adult patients. Am J Crit Care. 2006 Jul;15(4):420-7. PMID 16823021
- [Background] Geyer NM, Coetzee SK, Ellis SM, Uys LR. Relationship of nurses' intrapersonal characteristics with work performance and caring behaviors: A cross-sectional study. Nurs Health Sci. 2018 Sep;20(3):370-379. doi: 10.1111/nhs.12416. Epub 2018 Feb 28. PMID 29488674
- [Background] Guadagni V, Burles F, Ferrara M, Iaria G. The effects of sleep deprivation on emotional empathy. J Sleep Res. 2014 Dec;23(6):657-663. doi: 10.1111/jsr.12192. Epub 2014 Aug 13. PMID 25117004
- [Background] Hirsh AT, Jensen MP, Robinson ME. Evaluation of nurses' self-insight into their pain assessment and treatment decisions. J Pain. 2010 May;11(5):454-61. doi: 10.1016/j.jpain.2009.09.004. Epub 2009 Dec 16. PMID 20015702
- [Background] Hojat, M. (2016). Empathy in health professions education and patient care.
- [Background] Killgore WDS, Balkin TJ, Yarnell AM, Capaldi VF 2nd. Sleep deprivation impairs recognition of specific emotions. Neurobiol Sleep Circadian Rhythms. 2017 Jan 21;3:10-16. doi: 10.1016/j.nbscr.2017.01.001. eCollection 2017 Jun. PMID 31236499
- [Background] Kozlowski D, Hutchinson M, Hurley J, Rowley J, Sutherland J. The role of emotion in clinical decision making: an integrative literature review. BMC Med Educ. 2017 Dec 15;17(1):255. doi: 10.1186/s12909-017-1089-7. PMID 29246213
- [Background] Kyle SD, Beattie L, Spiegelhalder K, Rogers Z, Espie CA. Altered emotion perception in insomnia disorder. Sleep. 2014 Apr 1;37(4):775-83. doi: 10.5665/sleep.3588. PMID 24899765
- [Background] Kang Y, Moyle W, Venturato L. Korean nurses' attitudes towards older people with dementia in acute care settings. Int J Older People Nurs. 2011 Jun;6(2):143-52. doi: 10.1111/j.1748-3743.2010.00254.x. Epub 2010 Oct 28. PMID 21539719
- [Background] Mercer SW, Reynolds WJ. Empathy and quality of care. Br J Gen Pract. 2002 Oct;52 Suppl(Suppl):S9-12. PMID 12389763
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Owens JA. Sleep loss and fatigue in healthcare professionals. J Perinat Neonatal Nurs. 2007 Apr-Jun;21(2):92-100; quiz 101-2. doi: 10.1097/01.JPN.0000270624.64584.9d. PMID 17505227
- [Background] Rosen IM, Gimotty PA, Shea JA, Bellini LM. Evolution of sleep quantity, sleep deprivation, mood disturbances, empathy, and burnout among interns. Acad Med. 2006 Jan;81(1):82-5. doi: 10.1097/00001888-200601000-00020. PMID 16377826
- [Background] Sampson FC, Goodacre SW, O'Cathain A. The Reality of Pain Scoring in the Emergency Department: Findings From a Multiple Case Study Design. Ann Emerg Med. 2019 Oct;74(4):538-548. doi: 10.1016/j.annemergmed.2019.02.018. Epub 2019 Apr 5. PMID 30955987
- [Background] Tempesta D, Socci V, De Gennaro L, Ferrara M. Sleep and emotional processing. Sleep Med Rev. 2018 Aug;40:183-195. doi: 10.1016/j.smrv.2017.12.005. Epub 2017 Dec 22. PMID 29395984